CLINICAL TRIAL: NCT04826081
Title: Prospective Study on the Risks of Symptomatic Dengue on Pregnancy
Brief Title: Study on the Risks of Symptomatic Dengue on Pregnancy
Acronym: ERiDenG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/CHU/41
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Dengue; Pregnancy
Keywords: dengue fever ; pregnancy
MeSH Terms: conditions — Dengue | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: women who contracted symptomatic dengue fever during pregnancy
  Interventions: Other: data collection
- Control: women who did not contract symptomatic dengue fever during pregnancy
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
Dengue fever is the most common arbovirus worldwide (390 million people infected per year) and is a global public health problem. This public health problem is also becoming European due to its rapid expansion over the past decade with an increase in cases of 400% and the appearance of the first indigenous cases of dengue in Europe. Studies on the consequences of dengue fever on pregnancy find contradictory results. In fact, most of these studies are observational studies describing the risk of dengue fever for pregnancy, without comparison with a control group or comparing the different pregnancy morbidities to those found during pregnancy in the general population. Other research is retrospective case-control studies with major biases in the definitions of obstetric complications, which makes the results questionable.

The study therefore proposes to carry out a prospective case-control study with rigorous matching criteria, strict definitions of cases, controls and obstetric complications.

ELIGIBILITY:
Inclusion Criteria for the case :

* Pregnant patients
* Major
* Affiliated with social security
* Symptomatic or pauci-symptomatic dengue
* Biological confirmation of dengue fever

Inclusion Criteria for the control :

* Pregnant patients
* Major
* Affiliated with social security
* Asymptomatic

Exclusion Criteria for the 2 group :

* Multiple pregnancy
* Patient's refusal
* Protected persons: person deprived of liberty by judicial or administrative decision, minor, and person subject to a legal protection measure: guardianship or curators)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case : Patients who contracted dengue fever during pregnancy Control : Patient who does not get dengue fever during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the difference in the proportion of intrauterine growth retardation (IUGR) between the Case group and the Control group | at childbirth
  Birth weight <3rd percentile according to Sentinel Network Perinatal Database : AUDIPOG

SECONDARY OUTCOMES:
Evaluate the difference in the proportion of prematurity between the case group and the control group | at childbirth
  Prematurity: birth between 22 and 37 weeks of amenorrhea
Evaluate the difference in the proportion of late miscarriage between the case group and the control group | at childbirth
  late miscarriage: Birth between 14 and 22 weeks of amenorrhea
Evaluate the difference in the proportion of fetal death in utero between the case group and the control group | at childbirth
  fetal death in utero : Negative cardiac activity in utero between 14 weeks and before childbirth
Evaluate the difference in the proportion of preeclampsia between the case group and the control group | at childbirth
  preeclampsia: Arterial hypertension> 140 and / or 90 mmHg and proteinuria / 24h> 0.3g / 24h
Evaluate the difference in the proportion of bleeding from delivery between the case group and the control group between the case group and the control group | at childbirth
  bleeding from delivery: Blood loss> 500 mL in immediate postpartum up to 2 hours postpartum
Evaluate the difference in the proportion of small weight for gestational age between the case group and the control group between the case group and the control group | at childbirth
  Birth weight <10th percentile according to Sentinel Network Perinatal Database : AUDIPOG

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No